CLINICAL TRIAL: NCT01220362
Title: Effects of Thoracic Epidural Analgesia and Surgery on Lower Urinary Tract Function: A Randomized, Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Dr. med. Patrick Wüthrich, Department of Anesthesiology and Pain Therapy,University Hospital Bern Inselspital Bern
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 093/10
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Analgesia, Epidural; Urodynamics; Urinary Retention
Keywords: Analgesia, Epidural; Urodynamics; Urinary Retention
MeSH Terms: conditions — Agnosia; Urinary Retention | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Other): Bupivacaine 0.125%
  Interventions: Drug: Bupivacain 0.125%
- Group 2 (Other): Bupivacaine 0.125%/Fentanyl 2mcg/ml
  Interventions: Drug: Bupivacain 0.125%/Fentanyl 2mcg/ml

INTERVENTIONS:
Drug: Bupivacain 0.125% — Bupivacain 0.125%
  Arms: Group 1
Drug: Bupivacain 0.125%/Fentanyl 2mcg/ml — Bupivacain 0.125%/Fentanyl 2mcg/ml
  Arms: Group 2

SUMMARY:
Postoperative urinary retention (POUR) is one of the most common complications after surgery and neuraxial anesthesia of which the treatment of choice is bladder catheterization 1. It has been a common practice to place an indwelling catheter in the bladder in patients receiving epidural analgesia and to leave the catheter as long as the epidural analgesia is maintained despite a lack of evidence supporting this approach.

Transurethral catheterization is associated with significant morbidity such as patient discomfort, urethral trauma and urinary tract infections (UTI). Prolonged catheterization is the primary risk factor for catheter associated UTI (CAUTI), which is one of the most common nosocomial infections and can prolong hospitalisation 2. For this reason there is a growing focus on limiting the duration of catheterization and finding methods to avoid unnecessary catheterization in perioperative medicine 3,4.

Lower urinary tract function depends on coordinated actions between the detrusor muscle and the external urethral sphincter. Motorneurons of both muscles are located in the sacral spinal cord between L1 and S4. Most afferent fibers from the bladder enter the sacral cord through the pelvic nerve at segments L4-S2.

Because epidural analgesia can be performed at various levels of the spinal cord, it is possible to block only a portion of the spinal cord (segmental blockade). Based on the innervation of the bladder and sphincter between L1 and S4 it can be assumed that epidural analgesia within segments T4-6 to T10-12 has no or minimal influence on lower urinary tract function.

In a previous study, we found, against our expectations that thoracic epidural analgesia (TEA) significantly inhibits the detrusor muscle during voiding, resulting in clinically relevant post-void residuals which required monitoring or catheterisation 5. Because the study adopted a before-after design, we could not definitively identify the mechanisms responsible for this change in bladder function. In particular, we could not determine whether TEA per se or surgery was the main cause. Concerning TEA, it remains unclear which compounds of the solution, the local anesthetic, the opioid or both are responsible for the observed changes in lower urinary tract function.

The aim of this study is to compare lower urinary tract function before and during TEA with two different epidural solutions (group 1: bupivacaine 1.25 mg/ml vs group 2: bupivacaine 1.25 mg/ml combined with fentanyl 2 µg/ml) within segments T4-6 to T10-12 for postoperative pain treatment in patients undergoing lumbotomy for open renal surgery.

We expect that a better understanding of lower urinary tract function during TEA could lead to a more restrictive use of indwelling transurethral catheters perioperatively.

DETAILED DESCRIPTION:
Background

Acute urinary retention is one of the most common complications after surgery and anesthesia. It can occur in patients of both sexes and all age groups and after all types of surgical procedures. It is linked to several factors including increased intravenous fluids, postoperative pain and type of anaesthesia 1.

Micturition depends on coordinated actions between the detrusor muscle and the external urethral sphincter. Motorneurons of both muscles are located in the sacral spinal cord and coordination between them occurs in the pontine tegmentum of the caudal brain stem. Motorneurons innervating the external urethral sphincter are located in the nucleus of Onuf, extending from segment S1 to S3. The detrusor smooth muscle is innervated by parasympathetic fibers, which reside in the sacral intermediolateral cell group and are located in S2-4. Sympathetic fibers innervating the bladder and urethra play an important role in promoting continence and are located in the intermediolateral cell group of the lumbar cord (L1-L4). Most afferent fibers from the bladder enter the sacral cord through the pelvic nerve at segments L4-S2 and the majority are thin myelinated or unmyelinated.

There are few studies on the urodynamic effects of various anaesthetic agents 2-8, which mainly focused on lumbar epidural anaesthesia. Under the influence of epidural analgesia, patients may not feel the sensation of bladder filling, which can result in urinary retention and bladder overdistension. Overfilling of the bladder can stretch and in some cases permanently damage the detrusor muscle.

Because epidural anesthesia can be performed at various levels of the spinal cord, it is possible to block only a portion of the spinal cord (segmental blockade). Based on knowledge of the bladder innervations, it can be assumed that epidural analgesia within segments T4-6 to T10-12 has no or minimal influences on lower urinary tract function.

In a previous study, we found, against our expectations that thoracic epidural analgesia significantly inhibits the detrusor muscle during voiding, resulting in clinically relevant post void residuals which required monitoring or transurethral catheterisation 9. Because the study adopted a before-after design, we could not definitively identify the mechanisms responsible for bladder dysfunction. In particular, we could not say whether thoracic epidural analgesia per se or surgery was the cause of bladder dysfunction. Furthermore, it remains which ingredients, whether the local anesthetic, the opioid or both are behind changes in voiding function.

Objective

In our previous studies, we found that TEA significantly inhibits the detrusor muscle during voiding, resulting in clinically relevant post-void residuals which required monitoring or catheterization with similar findings 5,30.

Because these studies adopted a before-after design, we could not definitively identify the mechanisms responsible for lower urinary tract dysfunction. In particular, we could not say whether TEA per se or surgery was the cause of lower urinary tract dysfunction. Furthermore, it remains unclear which compounds in the epidural solution, the local anesthetic, the opioid or both are behind the observed changes in lower urinary tract function.

The objectives of this study are to determine if TEA per se or surgery are the cause of bladder dysfunction and which drugs in the epidural solution are responsible for this effect.

Methods

Randomised controlled double-blind study. Patients will be randomly allocated to one of the two groups by a computer-generated randomization list. Randomization will be stratified by gender, in order to reach an equal number of male and females in the two groups. Patients and investigators will be blinded to the epidural solution administrated.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Open kidney surgery with lumbotomy
* Thoracic epidural analgesia
* International Prostate Symptom Score (IPSS) < 7
* Preoperative residual urine volume < 100ml

Exclusion Criteria

* Contraindications to epidural analgesia or refusal
* Preoperative residual urine volume > 100ml
* International Prostate Symptom Score (IPSS) > 7
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Difference in post-void residual between bupivacaine (group 1) and bupivacaine-fentanyl (group 2) after surgery on day 2 or 3, depending on patient mobilisation. | day 2 or 3 after surgery

SECONDARY OUTCOMES:
Difference in post-void residual before and after surgery under segmental blockade. | day 2 or 3 after surgery
Difference in secondary outcomes (see 2.1.2.) between group 1 and group 2 before surgery | day 2 or 3 after surgery
Difference in secondary outcomes (see 2.1.2.) before and after surgery under segmental blockade. | day 2 or 3 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Fiona C Burkhard, Prof, Study Chair — Dep. of urology, University Hospital Bern, 3010 Bern, Switzerland
Locations (1):
- Dep. of Anesthesiology and Pain Therapy, University Hospital Bern, 3010 Bern,Switzerland, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] Baldini G, Bagry H, Aprikian A, Carli F. Postoperative urinary retention: anesthetic and perioperative considerations. Anesthesiology. 2009 May;110(5):1139-57. doi: 10.1097/ALN.0b013e31819f7aea. PMID 19352147
- [Result] Wuethrich PY, Kessler TM, Panicker JN, Curatolo M, Burkhard FC. Detrusor activity is impaired during thoracic epidural analgesia after open renal surgery. Anesthesiology. 2010 Jun;112(6):1345-9. doi: 10.1097/ALN.0b013e3181d4f4fe. PMID 20461004